CLINICAL TRIAL: NCT00575666
Title: Intranasal Insulin Treatment in Patients With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other); Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Xiaoduo Fan, Principal Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007-P-000731
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Results first posted 2012-12-17 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-11

CONDITIONS: Schizophrenia
Keywords: cognition, psychopathology
MeSH Terms: conditions — Schizophrenia | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Intranasal Insulin Treatment
  Interventions: Drug: Insulin or Placebo
- B (Placebo Comparator): Drug: Placebo
  Interventions: Drug: Insulin or Placebo

INTERVENTIONS:
Drug: Insulin or Placebo — intranasal, 40IU, 4 times daily

SUMMARY:
This study is an 8-week, randomized, double-blind, placebo-controlled trial of intranasal insulin as an adjunctive therapy, with a 4-week follow-up, in 60 non-diabetic schizophrenia subjects to examine insulin's effect on psychopathology and cognition. In addition, the study will examine insulin's effects on weight, food intake, resting energy expenditure, and body composition.

DETAILED DESCRIPTION:
The specific aims include:

Primary aims

1. Examine the efficacy of intranasal regular insulin (40 IU 4 times per day) in improving cognitive deficits in patients with schizophrenia.
2. Examine the efficacy of intranasal regular insulin in improving negative symptoms and positive symptoms of schizophrenia.

Secondary aims

1. Examine intranasal insulin's effects on weight, food intake and resting energy expenditure.
2. Examine intranasal insulin's effects on body composition, waist circumference, and waist/hip ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years.
2. Diagnosis of schizophrenia, any subtype or schizoaffective disorder, any subtype.
3. Stable dose of the current antipsychotic drug for at least one month.
4. Well established compliance with outpatient treatment per treating clinician's judgement.
5. Able to complete the cognitive assessment battery (must be English speaking).
6. Female subjects will be eligible to participate in the study if they are of non-childbearing potential or of child-bearing potential and willing to practice appropriate birth control methods (complete abstinence from sexual intercourse, female sterilization, sterilization of male partner, implants of levonorgestrel, injectable progestogen, oral contraceptives, intrauterine devices, or double barrier methods of contraception using spermicide with either a condom or diaphragm) during the study.

Exclusion Criteria:

1. Inability to provide informed consent.
2. Current substance abuse.
3. Psychiatrically unstable per treating clinician's judgement.
4. Significant medical illnesses including uncontrolled hypertension, diabetes, seizure. disorder, severe cardiovascular, cerebrovascular, pulmonary, or thyroid diseases.
5. Pregnancy or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2007-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoduo Fan, MD, MPH, MS, Principal Investigator — UMass Medical School
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Freedom Trail Clinic at the Erich Lindemann Mental Health Center and were studied at the Massachusetts General Hospital Clinical Research Center (MGH CRC), Boston.
Pre-assignment Details: After providing written informed consent, subjects underwent a diagnostic evaluation by a research psychiatrist using the Structured Clinical Interview for DSM-IV (SCID). All subjects were screened and enrolled based on eligibility criteria. Baseline study assessments were completed prior to intervention.
Groups:
- Intervention: Insulin: Intranasal insulin treatment, daily dosage 160 IU insulin for 8 weeks with a 4 week follow-up
- Intervention: Placebo: Placebo group, daily dosage 160 IU placebo for 8 weeks with 4 week follow-up
Period: Overall Study
Arm/Group | Intervention: Insulin | Intervention: Placebo
Started | 21 | 24
Completed | 17 | 21
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention: Insulin | Intervention: Placebo | Total
Number analyzed (Participants) | 21 | 24 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 24 | 45
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 49.2 (9.3) | 43.8 (9.2) | 46.0 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 18 | 18 | 36
Region of Enrollment [Number; unit: participants]
  United States | 21 | 24 | 45

OUTCOME MEASURES:

1. Primary Outcome: Cognitive Function- Digit Span Total
Description: Subjects completed the digit span task. Assessment was completed at Screening/Baseline, Week 4, and Week 8. Higher scores represent higher recall accuracy, and therefore less advanced psychopathology. Min score= 0, Max score= 30. Week 8 values are displayed below.
Time Frame: Week 8
Population: All subjects who completed the study for each Arm/Group were analyzed on cognitive function measures; study completion allows for calculation of change scores.
Measure: Mean (Standard Deviation); unit: Items correct
Groups:
- Humulin; Placebo: 160 IU per day for 8 weeks
Arm/Group | Humulin | Placebo
Number analyzed (Participants) | 17 | 21
Items correct | 13.3 (4.0) | 14.1 (4.9)

2. Primary Outcome: Cognitive Function- Verbal Fluency
Description: Subjects completed a verbal fluency test. Assessment was completed at Screening/Baseline, Week 4, and Week 8. Higher scores represent higher levels of verbal fluency, and therefore less advanced psychopathology. Min score= 0, Max score= N/A. Week 8 values are displayed below.
Time Frame: Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Words correct
Arm/Group | Humulin | Placebo
Number analyzed (Participants) | 17 | 21
Words correct | 27.9 (11.6) | 28.0 (13.3)

3. Primary Outcome: Cognitive Function- HVLT Immediate Recall Total
Description: Subjects completed a word recall task. Assessment was completed at Screening/Baseline, Week 4, and Week 8. Higher scores represent higher recall accuracy, and therefore less advanced psychopathology. Min score= 0, Max score= 36. Week 8 values are displayed below.
Time Frame: Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Words correct
Arm/Group | Humulin | Placebo
Number analyzed (Participants) | 17 | 21
Words correct | 21.4 (8.4) | 23.6 (7.1)

4. Primary Outcome: Cognitive Function- HVLT Delayed Recall Total
Description: Subjects completed a delayed word recall task. Assessments were completed at Screening/Baseline, Week 4, and Week 8. Higher scores represent higher recall accuracy, and therefore less advanced psychopathology. Min score= 0, Max score= 12. Week 8 values are displayed below.
Time Frame: Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Words correct
Arm/Group | Humulin | Placebo
Number analyzed (Participants) | 17 | 21
Words correct | 6.8 (3.6) | 7.8 (3.2)

5. Primary Outcome: Cognitive Function- Trails A
Description: Subjects completed a timed "trails" (i.e. connect-the-dots) test. Assessments were completed at Screening/Baseline, Week 4, and Week 8. Scores were measured by time to complete in seconds. Max score= N/A. Lower values represent less advanced psychopathology. Week 8 values are displayed below.
Time Frame: Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Humulin | Placebo
Number analyzed (Participants) | 17 | 21
Seconds | 60.6 (35) | 52.3 (23.2)

6. Primary Outcome: Cognitive Function- Trails B
Description: Subjects completed a timed "trails" (i.e. connect the dots) test. Assessments were completed at Screening/Baseline, Week 4, and Week 8. Scores were mesured by time to complete in seconds. Max score= N/A. Lower values represent less advanced psychopathology. Week 8 values are displayed below.
Time Frame: Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Humulin | Placebo
Number analyzed (Participants) | 17 | 21
Seconds | 131.5 (62) | 118.6 (44.1)

7. Primary Outcome: Cognitive Function- CPT D Prime Score
Description: Subjects completed a computer-based cognitive test designed to measure sustained attention (attention to a specific stimulus over a period of several minutes) before and after intranasal treatment. During this test, participants respond as quickly as possible to any consecutive presentation of identical stimuli on the computer screen. The stimuli (2, 3, and 4-digit targets) were presented with increasing cognitive load in successive blocks. Correct responses, responses made to the second of 2 identical stimuli presented in a row, were scored as hits. False alarms were also recorded. The "d prime score" is a score given to each participant on a scale of 0.0- 1.0 in which discrimination sensitivity is measured. A score of zero equates to no sensitivity, whereas a score of 1.0 equates to perfect sensitivity. Values below represent postreatment performance minus pretreatment performance. Higher scores represent less advanced psychopathology. Week 8 values are displayed below.
Time Frame: Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: D prime score
Arm/Group | Humulin | Placebo
Number analyzed (Participants) | 17 | 21
D prime score | 1.9 (1) | 2.1 (1)

8. Primary Outcome: Cognitive Function- CPT Hits Rate (Proportion)
Description: Subjects completed a computer-based cognitive test. The test is described in detail in a previous outcome measure ("CPT d prime score"). Hits rate was defined as the proportion of correct responses to the relevant stimuli (response to two identical targets) compared to total responses (total hits). Assessments were completed at Screening/Baseline, Week 4, and Week 8. Hits rate as a proportion of total hits was measured. Min score= 0, Max score= 1.0. Higher values represent higher stimulus recognition accuracy, and thus less advanced psychopathology. Week 8 values are displayed below.
Time Frame: Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Proportion of total hits
Arm/Group | Humulin | Placebo
Number analyzed (Participants) | 17 | 21
Proportion of total hits | 0.7 (0.2) | 0.7 (0.2)

9. Primary Outcome: Cognitive Function- CPT Reaction Time of Hits (Milliseconds)
Description: Subjects completed a computer-based cognitive functioning test designed to measure sustained attention (attention to a stimulus over a period of several minutes). The test is described in detail in a previous outcome measure ("CPT d prime score"). Reaction time of hits is defined as the average time each participant took to respond correctly to relevant stimuli. Assessments were completed at Screening/Baseline, Week 4, and Week 8. Reaction time was measured in milliseconds. Max score= N/A. Lower values represent less advanced psychopathology. Week 8 values are displayed below.
Time Frame: Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Humulin | Placebo
Number analyzed (Participants) | 17 | 21
Milliseconds | 554.1 (109.4) | 552.9 (73.7)

10. Primary Outcome: Cognitive Function- CPT False-alarm Rate (Proportion)
Description: Subjects completed a computer-based cognitive functioning test designed to measure sustained attention (attention to a stimulus over a period of several minutes). False alarm rate is defined as the proportion of overall hits that were in response to an incorrect stimulus (two consecutive non-identical targets). Assessments were completed at Screening/Baseline, Week 4, and Week 8. False-alarm hits were measured as a proportion of total hits. Min score= 0, Max score= 1.0. Lower values represent higher hit accuracy and less advanced psychopathology. Week 8 values are displayed below.
Time Frame: Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Proportion of total hits
Arm/Group | Humulin | Placebo
Number analyzed (Participants) | 17 | 21
Proportion of total hits | 0.1 (0.1) | 0.1 (0.1)

11. Primary Outcome: Psychopathology- PANSS Total
Description: Positive symptoms, negative symptoms, and general psychopatholgy of schizophrenia were measured at Screening/Baseline, Week 4, and Week 8. The assessment consisted of 30 total items, with each item measured on a seven-point scale (1= absent, 4= moderate, 7= extreme). Min score= 30, Max score= 210. Higher scores represent more advanced psychopathology. Week 8 values are displayed below.
Time Frame: Week 8
Population: All subjects who completed the study for each Arm/Group were analyzed on psychopathology measures; study completion allows for calculation of change scores.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humulin | Placebo
Number analyzed (Participants) | 17 | 21
units on a scale | 74.3 (19.5) | 74.1 (13.5)

12. Primary Outcome: Psychopathology- PANSS Positive
Description: Positive symptoms of schizophrenia were measured at Screening/Baseline, Week 4, and Week 8. The assessment consisted of seven items, with each item measured on a seven-point scale (1= absent, 4= moderate, 7= extreme). Min score= 7, Max score= 49. Higher scores represent more advanced psychopathology. Week 8 values are displayed below.
Time Frame: Week 8
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humulin | Placebo
Number analyzed (Participants) | 17 | 21
units on a scale | 17.2 (5.6) | 16.8 (5.1)

13. Primary Outcome: Psychopathology- PANSS Negative
Description: Negative symptoms of schizophrenia were measured at Screening/Baseline, Week 4, and Week 8. Assessment consisted of seven-items, with each item measured on a seven-point scale (1= absent, 4= moderate, 7= extreme). Min score= 7, Max score= 49. Higher scores represent more advanced psychopathology. Week 8 values are displayed below.
Time Frame: Week 8
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humulin | Placebo
Number analyzed (Participants) | 17 | 21
units on a scale | 20.8 (6.0) | 20.7 (5.8)

14. Primary Outcome: Psychopathology- PANSS General Psychopathology
Description: General psychopathology was measured at Screening/Baseline, Week 4, and Week 8. The assessment consisted of 16 items, with each item measured on a seven-point scale (1= absent, 4= moderate, 7= extreme). Min score= 16, Max score= 112. Higher scores represent more advanced psychopathology. Week 8 values are displayed below.
Time Frame: Week 8
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humulin | Placebo
Number analyzed (Participants) | 17 | 21
units on a scale | 36.3 (9.9) | 36.6 (7.4)

15. Primary Outcome: Psychopathology- SANS Total
Description: Negative symptoms of schizophrenia were measured at Screening/Baseline, Week 4, and Week 8. Assessment consisted of 25 items, with each item measured on a six-point scale (0= none, 3= moderate, 5= severe). Min score= 0, Max score= 125. Higher scores represent more advanced psychopathology. Week 8 values are displayed below.
Time Frame: Week 8
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humulin | Placebo
Number analyzed (Participants) | 17 | 21
units on a scale | 30.8 (15.2) | 33.5 (14.3)

16. Primary Outcome: Psychopathology- CDSS Total
Description: Symptoms of depression were measured at Screening/Baseline, Week 4, and Week 8. Assessment consisted of 9 items, with each item measured on a four-point scale (0= absent, 3= severe). Min score= 0, Max score= 27. Higher scores represent more advanced psychopathology. Week 8 values are displayed below.
Time Frame: Week 8
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humulin | Placebo
Number analyzed (Participants) | 17 | 21
units on a scale | 2.1 (3.2) | 2.7 (4.4)

17. Primary Outcome: Psychopathology- QLS Total
Description: Quality of life was measured at Screening/Baseline, Week 4, and Week 8. Assessment consisted of 21 items, with each item measured on a seven-point scale (0= not present, 3= sometimes present, 6= always present). Min score= 0, Max score= 126. Higher scores represent lower quality of life. Week 8 values are displayed below.
Time Frame: Week 8
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humulin | Placebo
Number analyzed (Participants) | 17 | 21
units on a scale | 70.9 (16.3) | 67 (16.8)

ADVERSE EVENTS:
Time Frame: Data was monitored for potential SAEs and AEs for a period of 34 months. For each individual subject, the timeframe for SAE and AE reporting was 12 weeks.
Arm/Group | Intervention: Insulin | Intervention: Placebo
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/24
Other Adverse Events (participants affected / at risk) | 0/21 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes